CLINICAL TRIAL: NCT00306046
Title: Use of 18F-Fluoride Positron Emission Tomography in the Assessment and Evaluation of Therapy in Monostotic Paget's Disease of Bone
Brief Title: 18F-Fluoride Positron Emission Tomography (PET) in Paget's Disease of Bone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3.4528.03 F
Record Dates: First submitted 2006-03-20; First posted 2006-03-22 (Estimated); Last update posted 2006-03-22 (Estimated); Status verified 2006-03

CONDITIONS: Paget's Disease of Bone
Keywords: PETScan; Positron-Emission Tomography; Bisphosphonate; Biochemical Markers; Paget's Disease of Bone (monostotic and polyostotic)
MeSH Terms: conditions — Osteitis Deformans

INTERVENTIONS:
Drug: Bisphosphonate treatment

SUMMARY:
18 F-fluoride Positron emission tomography (PET) is able to demonstrate and quantify the metabolic activity locally in the skeleton (1). This technique should, therefore, also be able to demonstrate a dramatic decrease in the metabolic activity in localized monostotic Paget's disease lesions after therapy. In this condition, indeed, the usual biological markers may be unhelpful to assess the efficacy of therapy, because they are usually comprised in the normal range for single pagetic localizations, even before therapy (2). The main purpose of this trial is to assess the early and long term response of pagetic bone to bisphosphonate therapy.

DETAILED DESCRIPTION:
I. Background of the subject:

Paget's disease of bone is a condition characterized by a focal exuberant increase in bone remodeling, resulting in a number of important architectural abnormalities, potentially leading to bone deformity and bone fragility. This condition may be polyostotic or monostotic. Biological markers of bone remodeling, mainly alkaline phosphatase and markers of bone resorption such as urinary hydroxyproline, are commonly utilized to assess Paget's disease activity.

However, a monostotic Paget's disease is most frequently accompanied by biological markers still in the normal range (1). Conventional 99mTc MDP bone scan is able to localize the lesion. However, the changes observed with this technique after therapy and when the disease recurs do not help much to guide the clinician (3). Indeed, there can be some improvement on the conventional bone scans whereas on the X-ray films, worsening of the pagetic lesions might simultaneously be observed (4). The recurrence of the condition could also be missed by conventional bone scans (4). Therefore, PET scan using 18 Fluoride should by its metabolic approach be able to demonstrate the local activity of Paget's disease, to assess the efficacy of active drugs and to evidence the local recurrence of the disease, better than the conventional existing techniques.

II. Experimental approach and methods

1. 20 patients suffering from a Paget's disease of bone (polyostotic: n = 6; monostotic: n = 14) will be studied prior to and after 1, 6, and 12 months of bisphosphonate therapy. The polyostotic cases will serve to the preliminary feasibility study. A localized Paget's disease will include isolated Pagetic lesions in bones of the face and or the skull, the spine and of the (lower or upper) limbs.
2. Paget's disease confirmed by X rays will be quantified by biological parameters of bone remodeling: total alkaline phosphatase, bone specific alkaline phosphatase, serum C-telopeptide (CTX), urinary NTx corrected by creatinine in a morning spot urine after an overnight fast.
3. Routine biological parameters such as creatinine, full blood count, serum calcium, phosphate and magnesium, as well as 25OH vitamin D, 1,25(OH)2 vitamin D and iPTH will also be performed at the start and after therapy. A total duration of 5 years should be considered for the completion of the whole study. 18 Fluoride will be produced by the cyclotron, localized in Louvain-la-Neuve (Belgium).

   18F-fluoride is produced by the 18O(p,n) 18F nuclear reaction by bombarding an enriched H218O target with protons. 185 Mbq 18F will be injected.
4. Scans will be performed on a Siemens ECAT HR+ PET scanner. This machine consists of 32 rings of BGO (bismuth germanium oxide) detectors (40.5x43.9x30 mm size) yielding 63 transverse slices (2.425 mm thickness) in a 16.2 cm axial FOV. In 2D mode, the resolution of the HR+ scanner is typically 5.4 mm and 5.0 mm FWHM at 10 cm in the transaxial and axial directions, respectively. A dynamic acquisition centered on pagetic bones will be performed over 60 minutes, starting immediately at tracer injection. Data will be reconstructed by filtered backprojection and iterative methods, with attenuation correction obtained from a transmission scan performed before tracer injection. Dynamic acquisition will allow us to modelize the tracer uptake and calculate the influx constants by means of multi-compartmental analysis. Kinetic modeling has been shown to better discriminate between normal, osteoporotic and Pagetic bones (Cook et al, SNM 2001, Toronto) and we assume that small changes in bone metabolism during therapy will be more precisely assessed by kinetic modeling than by simple semi-quantitative indexes such as standardized uptake values (SUV). Nevertheless, we will prospectively compare different models and SUV measurements to further identify the most appropriate quantification method.

Effective radiation dose equivalent is 0.027 mSv/Mbq 18F-fluoride. Target organ is the urinary bladder wall (due to the urinary excretion of the unbound fraction of the tracer) with an estimated radiation dose of 0.25 mGy/MBq.

III. References

1. Cook GJ, Lodge MA, Blake GM, Marsden PK, Fogelman I. Differences in skeletal kinetics between vertebral and humeral bone measured by 18 F-fluoride positron emission tomography in postmenopausal women. J Bone Miner Res 2000; 15: 763-769.
2. Kanis JA, Gray RES. Long-term follow-up observations on treatment in Paget's disease of bone. Clin Orthop 1987; 217: 99-125.
3. Smith ML, Fogelman I, Ralston S et al. Correlation of skeletal uptake of 99mTc-diphosphonate and alkaline phosphatase before and after oral diphosphonate therapy in Paget's disease. Metab Bone Dis Relat Res 1984; 5: 167-170.
4. Merrick MV, Merrick JM. Observations on the natural history of Paget's disease. Clin Radiol 1985; 36: 169-174.
5. Vellenga CLJR, Pauwels EKJ, Bijvoet OLM et al. Scintigraphic aspects of the recurrence of treated Paget's disease of bone. J Nucl Med 1985; 54: 273-281.
6. A. Nzeusseu Toukap, M. Lonneux, J. Installe, A. Bolle, G. Depresseux, J.P. Devogelaer.

International Symposium of the National Association for the Relief of Paget's Disease. St Catherine's college, 17-18 july 2003, Oxford, UK.

18F-Fluoride Positron Emission Tomography : Preliminary assessment of therapy in Paget's Disease of Bone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a monostotic form of PDB (as attested by plain X-rays and 99mTc MDP bone scintigraphy)
* Bone pain linked to Paget's disease itself

Exclusion Criteria:

* Bisphosphonate therapy within the year prior to the study

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2002-02; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Adrien T. NZEUSSEU, MD, Principal Investigator — Université Catholique de Louvain; Max LONNEUX, MD, PhD, Principal Investigator — Université Catholique de Louvain; Johanne INSTALLE, MD, Principal Investigator — Université Catholique de Louvain; Anne BOL, PhD, Principal Investigator — Université Catholique de Louvain; Geneviève DEPRESSEUX, Principal Investigator — Université Catholique de Louvain; Jean-Pierre DEVOGELAER, MD, Study Director — Université Catholique de Louvain
Locations (1):
- Rheumatology, Molecular Imaging and Experimental Radiotherapy departments, Saint-Luc University Hospital, Catholic University of Louvain, Brussels, Belgium

REFERENCES:
- [Background] Installe J, Nzeusseu A, Bol A, Depresseux G, Devogelaer JP, Lonneux M. (18)F-fluoride PET for monitoring therapeutic response in Paget's disease of bone. J Nucl Med. 2005 Oct;46(10):1650-8. PMID 16204715